CLINICAL TRIAL: NCT04543461
Title: The American Lung Association (ALA) Lung Health Cohort
Brief Title: American Lung Association (ALA) Lung Health Cohort
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Lung Association (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00236497; U01HL146408 (NIH)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Diseases
Keywords: lung health; environmental exposure; chest CT; spirometry; biomarkers
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, urine, nasal curettage, nasosorption strips
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ALA-LHC is a longitudinal, multi-center cohort study that will enroll approximately 4,000 young adults between the ages of 25-35 who do not have severe lung disease. The overarching objective of the ALA-LHC is to establish a national cohort of young adults for the purpose of defining lung health and developing targets to intercept chronic lung disease at its earliest stages.

DETAILED DESCRIPTION:
The scientific goal of the study is to establish the relationship between a variety of factors (lifetime environmental exposures, fitness and physical activity, biomarkers, nasal respiratory epithelial transcriptome) and ideal versus impaired peak lung health (reserve and markers of susceptibility in investigators' model) in young adulthood. In addition to the initial baseline assessment, remote contacts (e.g., via text message, email, mail, or phone) at regular intervals will allow for both the retention of the participants as well as the collection of additional short-term follow-up information, i.e., within 4.5 years of enrollment. If additional funding becomes available, investigators will extend the study for an additional period of time to study factors related to long-term changes in lung health over time, i.e., at 5 years and beyond. Recruitment of participants will be conducted by the participating study sites along with national and regional efforts from the American Lung Association. Recruitment efforts will be supported by the study web site www.lung.org/lung-study

ELIGIBILITY:
Inclusion Criteria:

1- Age 25-35 years at the time of the baseline examination 2- Able to read and understand English or Spanish 3 -Has a social security number 4- Resident (citizen or non-citizen) of the United States (US) for at least 12 months prior to examination. Note: Individuals who are residents of the US who have temporarily spent time living outside of the US during the last 12 months (e.g., student exchange program, military posting) are eligible for participation.

5- Willing to provide contact information for at least 2 proxies who are likely to know the whereabouts and vital status of the participant

Exclusion Criteria:

1. Severe asthma, which is defined as any of the following:

   1. Current (i.e. at the time of the visit) GINA Step 4 or higher therapy (medium dose ICS/LABA or high dose ICS or add-on LAMA; Medium dose = >250 fluticasone, propionate =100 fluticasone furoate, >200 beclomethasone, >400 budesonide, >220 mometasone). We will accept low-dose ICS/LABA or medium dose ICS.

      OR
   2. 3 or more unscheduled healthcare visits (provider/urgent care/ER) for asthma in the past 12 months OR
   3. One asthma hospitalization in the past 12 months
2. History of any chronic lung disease other than asthma including but not limited to COPD, cystic fibrosis, pulmonary fibrosis, pulmonary hypertension
3. Current pregnancy
4. History of cancer other than non-melanoma skin cancer
5. Diagnosed cardiovascular diseases (i.e., congenital heart disease, coronary heart disease)
6. Inability to comply with study procedures, including

   1. Inability or unwillingness to provide informed consent
   2. Inability to perform study measurements
   3. Inability to be contacted by phone (via calls and/or text messaging) or email
7. Any condition in the opinion of the physician that puts the participant at risk by participating in the study (e.g., serious respiratory illness requiring antibiotics or steroids or severe fever at the time of the study visit).
8. Institutionalization

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults between 25 and 35 year of age at baseline
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pre-bronchodilator measurement of Forced Expiratory Volume in one second (FEV1) | Baseline
  Pre-bronchodilator measurements of FEV1 to determine bronchoconstriction. FEV1 is measured in liters of air. Severity of bronchoconstriction is based on predicted values published by National Health and Nutrition Examination Survey (NHANES III hankinson) for height, weight and age. Predicted values are reported as percent predicted with a result of 80% or greater considered normal
Pre-bronchodilator measurements of Forced Vital Capacity (FVC) | Baseline
  Pre-bronchodilator measurements FVC to determine lung volume. FVC is measured in liters of air. Participants predicted vital lung capacity is based on values published by National Health and Nutrition Examination Survey (NHANES III hankinson) for height, weight and age. Predicted values are reported as percent predicted with a result of 80% or greater considered normal

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kalhan, MD, Principal Investigator — Northwestern University
Locations (37):
- United States (37):
  - University Of Alabama, Birmingham, Alabama
  - University of Arizona-Tuscon, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Jacksonville, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush Universtiy, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - St. Vincent's Health System, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Medical College, Hawthorne, New York
  - New York University, New York, New York
  - Mt. Sinai, NYC, New York, New York
  - Columbia University, New York, New York
  - Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburg-Emphysema/COPD Research Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Vermont, Colchester, Vermont
  - University of Washington, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin